CLINICAL TRIAL: NCT06499051
Title: Epidemiology of Sexual Offenders. A Cross-sectional Study of Auvergne-Rhône-Alpes Referral Platforms
Brief Title: Epidemiology of French Sexual Offenders. A Cross-sectional Study
Acronym: ARAVS
Status: Recruiting | Type: Observational
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A01205-40
Record Dates: First submitted 2024-06-10; First posted 2024-07-12 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Psychiatric Disorder
Keywords: sexual offenses; epidemiology
MeSH Terms: conditions — Mental Disorders | interventions — Sex

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cognition, impulsivity, emotional regulation, sexuality, diagnosis, sexual violence, motivation, self-esteem, social desirability, and defense mechanisms — self-administered questionnaires

SUMMARY:
The epidemiology of sexual offenders has been poorly studied in the literature. A retrospective and prospective study will allow for the examination of the clinical profile of sexual offense perpetrators, risk and recurrence factors, as well as psychiatric or medical treatment. Since 2015, the Auvergne-Rhône-Alpes region has 8 reference platforms for sexual offense perpetrators, offering personalized assessment according to criteria defined by the Regional Health Agency (ARS). After this assessment, a multidisciplinary meeting is organized to define a tailored care plan. This study, called ARAVS (Auvergne Rhone-Alpes Sexual Offenders), aims to conduct an epidemiological, clinical, and socio-demographic study of patients in these platforms.

DETAILED DESCRIPTION:
The Auvergne-Rhône-Alpes region, prompted by the Regional Health Agency (ARS), established a unique system of reference platforms starting in 2015, covering a large part of the region's territory. These platforms aim to provide comprehensive care for sexual offense perpetrators in addition to the support provided by the CRIAVS (Resource Centers for Professionals Working with Sexual Offenders). There are currently 8 active reference platforms in the region: in Bourg-en Bresse (Ain), Roanne (Loire), Saint-Etienne (Loire), Lyon (Rhône), Clermont-Ferrand (Puy-de-Dôme), Grenoble (Isère), Annecy (Savoie), and Valence (Drôme).

Given this context, it seems pertinent to implement a retrospective-prospective study of the clinical and epidemiological characteristics of patients treated in these reference platforms to better understand this population. These results will contribute to a better understanding of sexual offense perpetrators in France, as there is limited large-scale clinical data available, and will help tailor care tools to the population being treated in the region. Standardizing the use of common tools, which are currently being used heterogeneously, will also enrich the resources available to clinicians across all platforms by generalizing their use.

The coordinated organization of the reference platform network in the Auvergne-Rhône-Alpes region constitutes a unique care network in France, conducive to a clinical analysis of patients and their care pathways. The project will thus allow for the study of care pathways, the clinical and social profile of sexual offenders, and the identification of risk factors for recurrence among patients based on the data collected.

ELIGIBILITY:
All sexual offenders who are part of the PFR and meet the inclusion criteria will be invited to participate in this study.

Inclusion criteria:

* Adults (age ≥ 18 years).
* Under injunction of care for a sexual offense.
* Or Awaiting sentencing for a sexual offense.
* Or Currently under legal proceedings for a sexual offense.
* Or Under a legal obligation for care related to a sexual offense.
* Or Falling within the scope of an alternative to incarceration for a sexual offense.

Exclusion criteria:

* Patient refusal to participate in the study.
* Patients with physical or mental incapacity to complete the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All sexual offenders who are part of the PFR and meet the inclusion criteria will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Risk of re-offending and associated factors of the participant | From May 2024 to May 2027
  Sexual offender recidivism risk will be assessed using Static99 scale. The Static-99 (Hanson & Thornton, 2000) is the most commonly used actuarial risk tool for estimating sexual offender recidivism risk.The risk assessment instrument Static-99R consists of ten items, where all but items 1 and 5 are dichotomous, resulting in 0 or 1 point being added to the total score. The total score, between -3 and 12, results in one out of five recommended risk levels: level I - very low risk (scores of -3 to -2), level II - below average risk (scores of -1 to 0), level III - average risk (scores of 1 to 3), level IVa - above average risk (scores of 4 to 5), and level IVb - well above average risk (scores of 6+).

SECONDARY OUTCOMES:
Impulsivity of the participant | From May 2024 to May 2027 (cross-sectional study)
  Impulsivity will be assessed using the UPPS-P ( Impulsive Behavior Scale) scale. Participants are asked to consider acts/incidents during the last 6 months when rating their behavior and attitudes on a 4-point scale, in which 1-Agree strongly, 2-Agree some, 3-Disagree some, 4-Disagree strongly. This is a 59-item scale measuring 5 impulsivity components: negative urgency, positive urgency, lack of premeditation, lack of perseverance, and sensation seeking.Scores are presented for each of five subscales, plus a total impulsivity score.In addition to the raw scores, the mean is calculated for the items on each subscale, from 1 to 4, where 1 indicates that the respondent did not endorse impulsive answers, and 4 indicates a high level of self-reported impulsivity.
Cognition of the participant | From May 2024 to May 2027 (cross-sectional study)
  Cognition will be assessed using The Patient Competency Rating Scale (PCRS). The PCRS consists of 30 items, each scored on a scale of 1 to 5, making the total score range from 30 to 150. The higher scores indicate greater competency in the list of skills on the test.
Emotional status of the participant | From May 2024 to May 2027 (cross-sectional study)
  Emotional status will be assessed using theTAS-20 (Toronto Alexithymia Scale) scale. The TAS-20 is a self-report scale that is comprised of 20 items. Items are rated using a 5-point Likert scale whereby 1 = strongly disagree and 5 = strongly agree. There are 5 items that are negatively keyed (items 4, 5, 10, 18 and 19). The total alexithymia score is the sum of responses to all 20 items.The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 = possible alexithymia.
Diagnosis of the participant | From May 2024 to May 2027 (cross-sectional study)
  Diagnosis will be assessed using the PCL-R scale (Psychopathy Checklist Revised). The scale includes 2 factors. Factor 1 is a measure of Emotional Detachment (e.g., superficial charm, manipulativeness, shallow affectivity, absence of guilt or empathy). Factor 2 is a measure of Antisocial Behavior (deviance from an early age, aggression, impulsivity, irresponsibility, proneness to boredom). There is also a total score. A total score of 10-19 diagnoses an individual as midly psychopathic. A score of 20-29 diagnoses them as moderately psychopathic. a score of 30-40 diagnoses them as severely psychopathic.
Cognitive distorsions of the participant | From May 2024 to May 2027 ((cross-sectional study)
  Cognitive distorsions will be assessed using the bumby RAPE (BRS) and MOLEST (BMS) scales. The MOLEST scale is composed of 38 items and the RAPE scale is composed of 36 items scored on a 4-point Likert scale from strongly agree to strongly disagree. The BMS consists of38 items with a range of total scores being a minimum of 38 and a maximum of 152, and the BRS consists of 36 items with a total score ranging from 36 to 144.
Pedophilic Interests of the participant | From May 2024 to May 2027 ((cross-sectional study)
  pedophilic interests will be assessed using the Revised Screening Scale for Pedophilic Interests (SSPI-2). The SSPI-2 score ranges from zero to five, with higher scores indicating sexual interest in children.
Motivation of the participant | From May 2024 to May 2027 ((cross-sectional study)
  Motivation will be assessed using the URICA (University of Rhode Island Change Assessment Scale) scale. This is is a 32 item self-report measure that includes 4 subscales measuring the stages of change: Precontemplation, Contemplation, Action, and Maintenance. Responses are given on a 5 point Likert scale ranging from (1=strong disagreement to 5=strong agreement), An overall readiness to change score is calculated using a weighted average of the four sub-scores, where 14 is the maximum possible score. A higher score corresponds to increased readiness to change
Self-esteem of the participant | From May 2024 to May 2027 (cross-sectional study)
  Self-esteem will be assessed using the Rosenberg scale. The scale ranges from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem.

CONTACTS AND LOCATIONS:
Locations (1):
- CRIAVS - Centre Hospitalier Le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No